CLINICAL TRIAL: NCT04288687
Title: PLATPARP: a Phase II Single-Arm Trial of Niraparib in Platinum-Sensitive Castration-Resistant Prostate Cancer with DNA Repair Defects
Brief Title: A Trial of Niraparib in Platinum-Sensitive Castration-Resistant Prostate Cancer with DNA Repair Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 21819
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib Arm (only arm) (Other): Niraparib 200 mg by mouth daily (2 x 100 mg pills) on a 28 day cycle
  Interventions: Drug: Niraparib Pill

INTERVENTIONS:
Drug: Niraparib Pill — Niraparib 200 mg by mouth daily (2 x 100 mg pills)

SUMMARY:
This study is designed to evaluate the initial safety and effectiveness of an investigational drug, niraparib, given to patients who have recently received platinum-based chemotherapy for the treatment of prostate cancer. The study enrolls participants with history of advanced prostate cancer that is growing despite standard hormonal therapies, such as androgen-deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma (mixed histology will be acceptable, but pure small cell histology is to be excluded).
2. ≥ 18 years of age.
3. No prior therapy with PARP inhibitor therapy.
4. Patients must have received at least 9 weeks of platinum-based chemotherapy for the treatment of mCRPC as the proximal treatment regimen prior to study screening. Patients must not have evidence of clinical or radiographic disease progression (per Investigator assessment) and should have adequately recovered from chemotherapy-related toxicities (at least 4 weeks following completion of chemotherapy, with treatment-related toxicities ≤ grade 1 per CTCAE version 5).
5. ECOG performance status of ≤ 2.
6. Documented evidence of a pathogenic or likely pathogenic DNA repair aberration in BRCA1/2, ATM, FANCA, PALB2, CHEK2, HDAC2, or BRIP1 through either somatic or germline testing from a CLIA certified laboratory.
7. Radiographic evidence for metastatic disease. Measureable disease (per RECIST) is not required for enrollment. (i.e. bone-only metastatic disease is permitted).
8. Patients with history of treated brain metastases are eligible if off systemic corticosteroids for at least 2 weeks.
9. Clinical evidence for castration-resistance, with total testosterone < 50 ng/dL. Patients who have not undergone bilateral orchiectomy must plan to continue ongoing androgen deprivation therapy for the duration of the trial therapy.
10. Patients must have adequate organ function, as confirmed by laboratory values obtained ≤ 14 calendar days prior to the first day of study therapy:

    Hematologic: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused)

    Hepatic: Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver). (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject may be eligible)

    Renal: Estimated creatinine clearance ≥ 45 mL/min using Cockcroft Gault formula.
11. Patients must have a projected life expectancy of at least 3 months.

Exclusion Criteria:

1. Prior therapy with a PARP inhibitor.
2. Presence of clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
3. Presence of known significant immunodeficiency, as determined by the treating investigator.
4. Presence of clinically significant active infections, as determined by the treating investigator.
5. Known allergy to niraparib or any of its components.
6. Prostate cancer with histologic evidence for pure small cell histology

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
rPFS6 | 6 months
  Assessment of the 6-month radiographic progression-free survival (rPFS) rate in patients with platinum-sensitive mCRPC harboring germline or somatic DNA repair defects as determined by Kaplan-Meier analysis.

SECONDARY OUTCOMES:
PSA30 | 3 months
  Proportion of patients achieving a ≥30% decline in PSA following the initiation of niraparib maintenance therapy
PSA50 | 3 months
  Proportion of patients achieving a ≥50% decline in PSA following the initiation of niraparib maintenance therapy
Time to PSA progression | 6 months
  Time until the first PSA increase that is >25% (and an absolute increase of ≥ 2 ng/ml) from the nadir PSA value following the initiation of niraparib maintenance therapy
Frequency and severity of adverse events (AEs) | 1 month
  Frequency and severity of adverse events (AEs), as assessed by CTCAE version 5.0, following the initiation of niraparib maintenance therapy
Overall survival (OS) | 12 months
  Time from start of study therapy to death due to any cause. Patients who are alive will be censored on the most recent date of patient contact

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Narayan, MD, Principal Investigator — Ambramson Cancer Center of the University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided